CLINICAL TRIAL: NCT02996292
Title: Assessment of Dentoalveolar Changes Resulting From Orthodontic Treatment of Crowding With Self-ligating Brackets Using CBCT Randomized Controlled Trial
Brief Title: Treatment of Crowding Without Extraction Using Self Ligating Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-19 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Crowding
Keywords: Crowding; Self ligating; CBCT; RCT
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Traditional brackets (Experimental): Fixed orthodontic appliances will be applied for aligning and leveling of teeth up to 19*25 stainless steel wires using traditional brackets; American Orthodontics Master® MBT 0.022" Brackets
  Interventions: Device: Traditional brackets
- Active self-ligating brackets (Experimental): Fixed orthodontic appliances will be applied for aligning and leveling of teeth up to 19*25 stainless steel wires using active self-ligating brackets; American orthodontics active self-ligating Empower® MBT 0.022"
  Interventions: Device: Active self-ligating brackets
- Passive self-ligating brackets (Experimental): Fixed orthodontic appliances will be applied for aligning and leveling of teeth up to 19*25 stainless steel wires using passive self-ligating brackets; American orthodontics passive self-ligating Empower® MBT 0.022"
  Interventions: Device: Passive self-ligating brackets

INTERVENTIONS:
Device: Traditional brackets — Treating of crowding using traditional brackets
  Arms: Traditional brackets
Device: Active self-ligating brackets — Treating of crowding using active self-ligating brackets
  Arms: Active self-ligating brackets
Device: Passive self-ligating brackets — Treating of crowding using passive self-ligating brackets
  Arms: Passive self-ligating brackets

SUMMARY:
This experimental study will evaluate the effect of active and passive self-ligating brackets in treatment of crowding, compared with the control group of conventional brackets in class I malocclusion without extraction.

The study sample will consist of 66 patients with 3-6mm crowding. The sample will be allocated randomly into two experimental groups, in addition to a control group.

The brackets will be applied using indirect bonding method for all patients. The dentoalveolar changes occurring after leveling and alignment teeth will be assessed by using CBCT radiographs; pre and post- treatment changes for each group will be evaluated individually.

DETAILED DESCRIPTION:
Producing of modern and various brackets systems both self- ligating and conventional make the 3 dimensional important in order to evaluate the root positions and to investigate EARR in multi root teeth, so the research will depend on CBCT to carry out these purposes in our study. Beside to compare the duration of alignment among groups.

Fixed appliances will be applied into three groups as 1. Active self ligating brackets (ASLB), 2. Passive self ligating brackets (PSLB), 3. Conventional brackets (CB) until reach to wire 19*25 S.S upper and lower. During leveling, thermal activated wires will be used in all patients.

CBCT images will be done before and after leveling and alignment of teeth to compare dentoalveolar changes between study groups.

ELIGIBILITY:
Inclusion Criteria:

* patients permanent dentition stage.
* crowding up to 6 mm
* Class I relationship.
* Good oral hygiene.

Exclusion Criteria:

* Poor oral hygiene.
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Class II or III skeletal anteroposterior relationship.
* Crowding less than 3mm and more than 6mm.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Speed of alignment | After 9 months
  Speed of alignment will be measured and compared between the groups.

SECONDARY OUTCOMES:
Changes of the torque and tipping of teeth | Evaluation before and after alignment and leveling teeth. (after 9 months)
  The torque and tipping of teeth will be evaluated before and after treatment and compared between the groups using CBCT images.
Changes of widths and depths of the dental arches | Evaluation before and after alignment and leveling teeth. (after 9 months)
  Changes of dental arches dimensions will be measured and compared between groups.
External apical root resorption | After 9 months
  External apical root resorption of each tooth on CBCT images (frequencies) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Burhan, PhD., Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be only available to the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Result] Badawi HM, Toogood RW, Carey JP, Heo G, Major PW. Torque expression of self-ligating brackets. Am J Orthod Dentofacial Orthop. 2008 May;133(5):721-8. doi: 10.1016/j.ajodo.2006.01.051. PMID 18456146
- [Result] Chan EK, Darendeliler MA, Petocz P, Jones AS. A new method for volumetric measurement of orthodontically induced root resorption craters. Eur J Oral Sci. 2004 Apr;112(2):134-9. doi: 10.1111/j.1600-0722.2004.00118.x. PMID 15056110
- [Result] Chen SS, Greenlee GM, Kim JE, Smith CL, Huang GJ. Systematic review of self-ligating brackets. Am J Orthod Dentofacial Orthop. 2010 Jun;137(6):726.e1-726.e18; discussion 726-7. doi: 10.1016/j.ajodo.2009.11.009. PMID 20685517
- [Result] Garcia-Figueroa MA, Raboud DW, Lam EW, Heo G, Major PW. Effect of buccolingual root angulation on the mesiodistal angulation shown on panoramic radiographs. Am J Orthod Dentofacial Orthop. 2008 Jul;134(1):93-9. doi: 10.1016/j.ajodo.2006.07.034. PMID 18617108
- [Result] Lagravere MO, Carey J, Toogood RW, Major PW. Three-dimensional accuracy of measurements made with software on cone-beam computed tomography images. Am J Orthod Dentofacial Orthop. 2008 Jul;134(1):112-6. doi: 10.1016/j.ajodo.2006.08.024. PMID 18617110
- [Result] Morina E, Eliades T, Pandis N, Jager A, Bourauel C. Torque expression of self-ligating brackets compared with conventional metallic, ceramic, and plastic brackets. Eur J Orthod. 2008 Jun;30(3):233-8. doi: 10.1093/ejo/cjn005. PMID 18540011
- [Result] Sifakakis I, Pandis N, Makou M, Eliades T, Bourauel C. A comparative assessment of the forces and moments generated at the maxillary incisors between conventional and self-ligating brackets using a reverse curve of Spee NiTi archwire. Aust Orthod J. 2010 Nov;26(2):127-33. PMID 21175021